CLINICAL TRIAL: NCT02492932
Title: The Second Try During Landmark Approach of the Internal Jugular Vein: an Ultrasonographic Prelocation Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CWJung_IJV
Record Dates: First submitted 2015-06-09; First posted 2015-07-09 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Jugular Veins
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IJV_2nd (Experimental): Ultrasonography examination of the patients who are assumed to take second attempt of internal jugular venous catheterization
  Interventions: Device: Ultrasonography

INTERVENTIONS:
Device: Ultrasonography — Ultrasonography evaluation of the internal jugular vein.

SUMMARY:
Two approaches are possible when the first finder needle attempt of the internal jugular vein cannulation fails; the needle can be turned slightly laterally or the puncture point can be moved slightly medially. This study is an ultrasonographic stimulation study to evaluate the success rate of turning the needle laterally and moving the puncture point medially, and to determine the proper angle or distance for the second try of internal jugular vein cannulation.

DETAILED DESCRIPTION:
Immediately after induction of general anesthesia, the patient's head is turned slightly, and the table is tilted at 10 degrees, and the puncture point estimated by the anatomical landmarks are marked on the patient's skin. The investigators obtain a sonographic view at the estimated puncture point. It is recorded "success" when the internal jugular vein is visualized on the ultrasonography, and the estimated needle path passes the internal jugular vein. It is recorded "failure" if the internal jugular vein is not visualized on the ultrasonography, and the estimated needle path does not pass the internal jugular vein. After "failure" of the first attempt, the probe is either turned laterally or moved medially until the internal jugular vein is visualized on the ultrasonography, and the estimated needle path passes the internal jugular vein. The angle and distance is recorded. The location of the carotid artery is always marked on the ultrasonography for evaluation of complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for general anesthesia

Exclusion Criteria:

* Refusal of consent
* Patients with C-spine injuries
* Patients with atlanto-axial instability
* Patients at risk of increased intracranial pressure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Success rate of internal jugular vein cannulation at the second attempt after failure of first attempt on ultrasonographic simulation | intraoperative

SECONDARY OUTCOMES:
Degree of lateral rotation or medial movement for successful puncture of second attemp | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea